CLINICAL TRIAL: NCT04143698
Title: Randomized Trial Comparing Reusable and Disposable Duodenoscopes for ERCP
Brief Title: Reusable Versus Disposable Duodenoscopes for ERCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1388902
Record Dates: First submitted 2019-06-05; First posted 2019-10-29 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Endoscopic Retrograde Cholangiopancreatography
Keywords: duodenoscopes; ERCP
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Disposable (single-use) duodenoscope (Active Comparator): This group will be using the disposable (single-use) duodenoscope during endoscopic retrograde cholangiopancreatography (ERCP).
  Interventions: Device: endoscopic retrograde cholangiopancreatography
- Reusable duodenoscope (Active Comparator): This group will be using the reusable duodenoscope during endoscopic retrograde cholangiopancreatography (ERCP).
  Interventions: Device: endoscopic retrograde cholangiopancreatography

INTERVENTIONS:
Device: endoscopic retrograde cholangiopancreatography — The duodenoscope will be passed to the duodenum in the standard fashion. Once the papilla has been identified in the duodenum, cannulation of the desired duct will be performed in the standard fashion, with the type of accessories used left to the discretion of the individual endoscopist performing the procedure. If cannulation is considered difficult, advanced cannulation techniques can be used per standard of care at the discretion of the individual endoscopist. The types of accessories used will be left to the discretion of the individual endoscopist and will be dependent on procedure indication and personal preference. Cross-over to the alternate duodenoscope type can be performed at any time if the desired technical maneuver cannot be performed with the designated duodenoscope.
  Other Names: ERCP

SUMMARY:
The aim of this randomized trial is to evaluate the technical aspects of disposable duodenoscopes and to compare the technical outcomes between the disposable (single-use) and reusable duodenoscopes.

DETAILED DESCRIPTION:
Given the recent reports on infection outbreaks, including carbapenem-resistant Enterobacteriaceae (CRE), caused by contaminated duodenoscopes used at endoscopic retrograde cholangiopancreatography (ERCP), a disposable (single-use) duodenoscope (Exalt, Single-Use Duodenoscope, Boston Scientific Corporation, Natick, MA) has been developed to circumvent this issue. However, there are currently no data on the technical features and outcomes of disposable duodenoscopes, in comparison with reusable duodenoscopes.

The aim of this randomized trial is therefore to evaluate the technical aspects of disposable duodenoscopes and to compare the technical outcomes between the two duodenoscope types.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Patients with native papilla
3. Requiring an ERCP procedure for biliary or pancreatic duct disorder, based on clinical symptoms and radiological findings at computed tomography or magnetic resonance cholangiopancreatography

Exclusion Criteria:

1. Age <18 years old
2. Unable to obtain informed consent
3. Pregnancy
4. Altered upper gastrointestinal surgical anatomy
5. Patients with percutaneous transhepatic biliary drainage catheters
6. Prior history of ERCP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-05-06 (Actual)

PRIMARY OUTCOMES:
Cannulation | 1 day
  The ease of cannulation of the desired duct (biliary or pancreatic), as measured by the total number of cannulation attempts to achieve successful cannulation of the desired duct.

SECONDARY OUTCOMES:
Ease of passage of duodenoscope and imaging and mechanical function of the duodenoscope | 1 day
  Ease of maneuverability of the duodenoscope to reach the major papilla, the imaging and mechanical function of the duodenoscope, measured on a five point scale with 1 being the easiest and 5 being the most difficult.
Ease of completion of interventions | 1 day
  Ease of completion of each step of the ERCP procedure, measured on a 5 point scale with 1 being the easiest and 5 being the most difficult.
Rate of use of advanced cannulation techniques | 1 day
  Need for use of advanced cannulation techniques
Rate of cross-over | 1 day
  Rate of cross-over to the alternate duodenoscope for completion of the procedure
Time taken for cannulation | 1 day
  Time taken for cannulation
Total duration of the procedure | 1 day
  Total duration of the procedure
Rate of adverse events | 7 days and 30 days
  Assessment of AEs and SAEs

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Varadarajulu, MD, Principal Investigator — AdventHealth Orlando
Locations (1):
- AdventHealth Orlando, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rauwers AW, Voor In 't Holt AF, Buijs JG, de Groot W, Hansen BE, Bruno MJ, Vos MC. High prevalence rate of digestive tract bacteria in duodenoscopes: a nationwide study. Gut. 2018 Sep;67(9):1637-1645. doi: 10.1136/gutjnl-2017-315082. Epub 2018 Apr 10. PMID 29636382
- [Background] Kim S, Russell D, Mohamadnejad M, Makker J, Sedarat A, Watson RR, Yang S, Hemarajata P, Humphries R, Rubin Z, Muthusamy VR. Risk factors associated with the transmission of carbapenem-resistant Enterobacteriaceae via contaminated duodenoscopes. Gastrointest Endosc. 2016 Jun;83(6):1121-9. doi: 10.1016/j.gie.2016.03.790. Epub 2016 Mar 16. PMID 26993149
- [Background] Alrabaa SF, Nguyen P, Sanderson R, Baluch A, Sandin RL, Kelker D, Karlapalem C, Thompson P, Sams K, Martin S, Montero J, Greene JN. Early identification and control of carbapenemase-producing Klebsiella pneumoniae, originating from contaminated endoscopic equipment. Am J Infect Control. 2013 Jun;41(6):562-4. doi: 10.1016/j.ajic.2012.07.008. Epub 2012 Nov 18. PMID 23171594
- [Background] Epstein L, Hunter JC, Arwady MA, Tsai V, Stein L, Gribogiannis M, Frias M, Guh AY, Laufer AS, Black S, Pacilli M, Moulton-Meissner H, Rasheed JK, Avillan JJ, Kitchel B, Limbago BM, MacCannell D, Lonsway D, Noble-Wang J, Conway J, Conover C, Vernon M, Kallen AJ. New Delhi metallo-beta-lactamase-producing carbapenem-resistant Escherichia coli associated with exposure to duodenoscopes. JAMA. 2014 Oct 8;312(14):1447-55. doi: 10.1001/jama.2014.12720. PMID 25291580
- [Background] Cotton PB, Eisen G, Romagnuolo J, Vargo J, Baron T, Tarnasky P, Schutz S, Jacobson B, Bott C, Petersen B. Grading the complexity of endoscopic procedures: results of an ASGE working party. Gastrointest Endosc. 2011 May;73(5):868-74. doi: 10.1016/j.gie.2010.12.036. Epub 2011 Mar 5. PMID 21377673
- [Background] Sahar N, La Selva D, Gluck M, Gan SI, Irani S, Larsen M, Ross AS, Kozarek RA. The ASGE grading system for ERCP can predict success and complication rates in a tertiary referral hospital. Surg Endosc. 2019 Feb;33(2):448-453. doi: 10.1007/s00464-018-6317-7. Epub 2018 Jul 9. PMID 29987568
- [Background] Testoni PA, Mariani A, Aabakken L, Arvanitakis M, Bories E, Costamagna G, Deviere J, Dinis-Ribeiro M, Dumonceau JM, Giovannini M, Gyokeres T, Hafner M, Halttunen J, Hassan C, Lopes L, Papanikolaou IS, Tham TC, Tringali A, van Hooft J, Williams EJ. Papillary cannulation and sphincterotomy techniques at ERCP: European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2016 Jul;48(7):657-83. doi: 10.1055/s-0042-108641. Epub 2016 Jun 14. PMID 27299638
- [Background] Liao WC, Angsuwatcharakon P, Isayama H, Dhir V, Devereaux B, Khor CJ, Ponnudurai R, Lakhtakia S, Lee DK, Ratanachu-Ek T, Yasuda I, Dy FT, Ho SH, Makmun D, Liang HL, Draganov PV, Rerknimitr R, Wang HP. International consensus recommendations for difficult biliary access. Gastrointest Endosc. 2017 Feb;85(2):295-304. doi: 10.1016/j.gie.2016.09.037. Epub 2016 Oct 5. No abstract available. PMID 27720741
- [Background] Bassi M, Luigiano C, Ghersi S, Fabbri C, Gibiino G, Balzani L, Iabichino G, Tringali A, Manta R, Mutignani M, Cennamo V. A multicenter randomized trial comparing the use of touch versus no-touch guidewire technique for deep biliary cannulation: the TNT study. Gastrointest Endosc. 2018 Jan;87(1):196-201. doi: 10.1016/j.gie.2017.05.008. Epub 2017 May 18. PMID 28527615
- [Background] Hwang JC, Yoo BM, Yang MJ, Lee YK, Lee JY, Lim K, Noh CK, Cho HJ, Kim SS, Kim JH. A prospective randomized study of loop-tip versus straight-tip guidewire in wire-guided biliary cannulation. Surg Endosc. 2018 Apr;32(4):1708-1713. doi: 10.1007/s00464-017-5851-z. Epub 2017 Sep 15. PMID 28916891
- [Background] Bassan MS, Sundaralingam P, Fanning SB, Lau J, Menon J, Ong E, Rerknimitr R, Seo DW, Teo EK, Wang HP, Reddy DN, Goh KL, Bourke MJ. The impact of wire caliber on ERCP outcomes: a multicenter randomized controlled trial of 0.025-inch and 0.035-inch guidewires. Gastrointest Endosc. 2018 Jun;87(6):1454-1460. doi: 10.1016/j.gie.2017.11.037. Epub 2018 Jan 6. PMID 29317269
- [Background] Buxbaum J, Leonor P, Tung J, Lane C, Sahakian A, Laine L. Randomized Trial of Endoscopist-Controlled vs. Assistant-Controlled Wire-Guided Cannulation of the Bile Duct. Am J Gastroenterol. 2016 Dec;111(12):1841-1847. doi: 10.1038/ajg.2016.268. Epub 2016 Jul 5. PMID 27377519
- [Derived] Bang JY, Hawes R, Varadarajulu S. Equivalent performance of single-use and reusable duodenoscopes in a randomised trial. Gut. 2021 May;70(5):838-844. doi: 10.1136/gutjnl-2020-321836. Epub 2020 Sep 7. PMID 32895332